CLINICAL TRIAL: NCT02370914
Title: Concussion Testing: A Novel Non-invasive Concussion Detection Device
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21114
Record Dates: First submitted 2014-02-21; First posted 2015-02-25 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suspected Concussive Event (SCE): When a subject is suspected of a concussion, a Nautilus NeuroWaveTM System recording is obtained from the subject and the recording is evaluated by a Jan Medical concussion algorithm. The subject is declared concussed or not per the algorithm. This is compared to a Sport Concussion Assessment Tool (SCAT) test.
  Interventions: Device: Nautilus NeuroWaveTM System; Behavioral: SCAT
- Control: All subjects at the start of study have a baseline recording using the Nautilus NeuroWaveTM System. These subjects are enrolled into the study as non-concussed and these recordings serve as control recordings. Additionally, some subjects from this cohort will be recorded again at the end of the study to obtain end of season recordings. These results are compared to a Sport Concussion Assessment Tool (SCAT) test.
  Interventions: Device: Nautilus NeuroWaveTM System; Behavioral: SCAT

INTERVENTIONS:
Device: Nautilus NeuroWaveTM System — Recording of subjects with Nautilus NeuroWave diagnostic device
  Other Names: Jan Medical Nautilus NeuroWave
Behavioral: SCAT — A Neurocognitive evaluation of the patients to assess for concussion.
  Other Names: Sports Concussion Assessment Test, SCAT2

SUMMARY:
The purpose of this study is to establish and evaluate a distinctive signal for concussion.

DETAILED DESCRIPTION:
The purpose of this study is to establish a non-invasive objective measurement for the detection of concussions with the Jan Medical Device (JMD). The study will assess the ability of this device to demonstrate unique signals that correlate with concussions. The study will also test the athletes at baseline at rest and during exertion to determine if there is a difference in the signal from exertion alone. The JMD is a non-invasive band that is placed around the participants head. The JMD detects a unique pattern of signals based on displacement of the skull from changes in blood flow during individual heartbeats. The athletes will be tested longitudinally to assess to changes over time, in addition to changes after impact

ELIGIBILITY:
Inclusion Criteria:

* Junior Varsity and Varsity Players a local High School.

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Varsity high school football players at a local High School.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Auerbach, Principal Investigator — Stanford University
Locations (1):
- Los Altos High School, Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic Device - Nautilus NeuroWave: Nautilus NeuroWave diagnostic device. Recordings were evaluated by a Jan Medical concussion algorithm .
  Nautilus NeuroWaveTM System: Recording of subjects with Nautilus NeuroWave diagnostic device
Period: Overall Study
Arm/Group | Diagnostic Device - Nautilus NeuroWave
Started | 84
Completed | 82
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic Device - Nautilus NeuroWave
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.33)
Sex/Gender, Customized [Number; unit: participants]
  Males | 82
Region of Enrollment [Number; unit: participants]
  United States | 82
Sport Concussion Assessment Tool- Second Edition (SCAT 2) [Mean (Standard Deviation); unit: units on a scale] — SCAT2 was used to perform baseline testing in athletes before the football season began. Of these, 9 without a concussion during the season, elected to have another recording done at the end of the year. If an athlete sustained an impact and sideline physicians or trainers regarded the impact as a concussion, the athlete had a SCAT2 test performed and Jan Medical Device (JMD) testing.The scale is based on total symptoms and symptom severity score, with 0 being least severe and 132 being most severe. In other words, the higher the the score value, the worse the condition. Score range is 0-132.
  units on a scale | 82.5 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: A Measure Assessing the Sensitivity and Specificity Rate Based on the Nautilus Neurowave Data
Description: Sensitivity (also called the true positive rate) measures the proportion of concussed participants that are correctly identified as such by utilizing the information within the Nautilus Neurowave data. Specificity (also called the true negative rate) measures the proportion of non-concussed participants that are correctly identified as such by utilizing the information within the Nautilus Neurowave data
  The information that is evaluated from within this data is recognized through the computation of two parameters, R1 and R2. Both R1 and R2 are measured by computing the frequency spectrum using an FFT of the Neurowave data and computing a ratio of the signal intensities at specific higher frequencies against specific lower frequencies within that spectrum. Based on this computation, the recorded data is evaluated as coming from a concussed participant if R1 >= 1.0 and R2 >= 0.66 and is considered non-concussed otherwise.
Time Frame: Individual assessments were made within 2 days of recording
Population: Analysis population includes all participants. Some of these participants were were declared concussed by the physician in the team during the course of the season. All baseline recordings were treated as from non-concussed participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diagnostic Device - Nautilus NeuroWave
Number analyzed (Participants) | 82
percentage of participants
  Sensitivity | 77 [50 to 92]
  Specificity | 87 [78 to 93]

ADVERSE EVENTS:
Time Frame: assessed from enrollment (baseline recording at beginning of sports season) to end of follow-up (end of sports season at 5 months)
Arm/Group | Diagnostic Device - Nautilus NeuroWave
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

LIMITATIONS AND CAVEATS:
This is a pilot study only. Only 15 concussions were observed from a single gender teenage population from one high school football team over one season. Further data from a broader population is needed to confirm results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No